CLINICAL TRIAL: NCT00639587
Title: A Double-blind, Parallel, Active Comparator Controlled, Randomized Trial; Comparison of the Efficacy and Safety in Children With Perennial Allergic Rhinitis of Cetirizine Tablets Versus Ketotifen Dry Syrup
Brief Title: Efficacy and Safety of Cetirizine Tablets Versus Ketotifen Dry Syrup in Children With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Study Director, UCB
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A00275
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2009-09-04 (Estimated); Status verified 2009-09

CONDITIONS: Rhinitis, Allergic, Perennial
Keywords: Cetirizine; Zyrtec
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Ketotifen; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ketotifen — Ketotifen dry syrup 0.1%; 1 mg b.i.d.; for 2 weeks
Drug: Cetirizine — Cetirizine tablet; 10 mg o.d.; for 2 weeks and 5 mg b.i.d.; for 2 weeks

SUMMARY:
Ketotifen is an established antihistamine drug, widely used in pediatric clinical practice in Japan. The objective of the study was to compare the efficacy and safety of cetirizine hydrochloride versus ketotifen dry syrup on children 7 years and older with perennial allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* had at least one of the 3 symptoms: sneezing, nasal discharge or nasal congestion;
* severity of nasal symptoms was moderate to severe during the observation period;
* criteria for allergic etiology of the disease fulfilled, i.e., positive IgE antibody test and positive eosinophil count in nasal discharge.

Exclusion Criteria:

* history of hypersensitivity to the ingredients of cetirizine or ketotifen formulation or to hydroxyzine;
* history of drug hypersensitivity;
* history of convulsive disorder;
* vasomotor rhinitis or eosinophilic rhinitis;
* asthma requiring treatment with adrenocortical hormones;
* concomitant diseases which could impede the efficacy evaluation of the study drug;
* subjects in the ascending-dose phase of hyposensitization therapy or non-modular therapy and who had not received the maintenance dosage;
* pollen allergy;
* malignant neoplasm.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2002-08; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Total symptom score (TSS) (nasal symptom score [sneezing, nasal discharge, nasal congestion] and rhinoscopy results) Safety: adverse events and laboratory assessments | TSS: 2 weeks - Safety: 3 weeks

SECONDARY OUTCOMES:
Total 2 symptoms score (T2SS) (sneezing, nasal discharge) Global Improvement Rating | T2SS: 2 weeks - Global Improvement Rating: at the end of the 2-week-treatment period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1-877-822-9493 (UCB)